CLINICAL TRIAL: NCT03315052
Title: Budesonide in Liver Transplantation
Brief Title: Budesonide for Immunosuppression After Liver Transplantation to Reduce Side Effects
Acronym: BILT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Delay in IRB approval
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-7959
Record Dates: First submitted 2017-10-13; First posted 2017-10-19 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Acute Cellular Graft Rejection; Liver Transplant Rejection
Keywords: Graft loss; Renal failure; Infection; Diabetes; Hypertension
MeSH Terms: conditions — Renal Insufficiency; Infections; Diabetes Mellitus; Hypertension | interventions — Budesonide; Tacrolimus; Mycophenolic Acid; Prednisone

STUDY DESIGN:
Intervention Model Description: Comparison of standard immunosuppression to immunosuppression incorporating budesonide in place of prednisone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Budesonide treatment arm (Experimental): Patients treated with budesonide in place of prednisone as part of immunosuppressive regimen
  Interventions: Drug: Budesonide; Drug: Tacrolimus（FK506）; Drug: Mycophenolate Mofetil
- Standard immunosuppression arm (Active Comparator): Patients treated with standard immunosuppression after liver transplant
  Interventions: Drug: Tacrolimus（FK506）; Drug: Mycophenolate Mofetil; Drug: Prednisone

INTERVENTIONS:
Drug: Budesonide — Oral steroid with high first-pass metabolism in liver
  Other Names: Enterocort
  Arms: Budesonide treatment arm
Drug: Tacrolimus（FK506） — Calcineurin immunosuppressant
  Other Names: Prograf
Drug: Mycophenolate Mofetil — Immunosupressant
  Other Names: Cellcept
Drug: Prednisone — Immunosuppresant
  Arms: Standard immunosuppression arm

SUMMARY:
Our hypothesis is that budesonide will provide effective hepatic ISP that will replace prednisone and allow lower systemic drug levels of FK, thus reducing the steroid- and calcineurin-associated complications often observed in the OLT population. This study is intended to investigate the therapeutic potential of this ISP combination.

DETAILED DESCRIPTION:
This study will be a randomized, open-label non-inferiority trial to assess the efficacy, safety and tolerability of budesonide in combination with low-dose FK and standard-dose MMF as post-OLT ISP in comparison to standard ISP (S-ISP). Subjects will include OLT patients age 18 years and older receiving their first single-organ living- or deceased-donor liver transplant. Subjects must have post-operative recovery of graft function and be able to take oral medications before beginning treatment according to the study protocol.

Subjects will be randomized to receive either (1) investigational oral ISP including budesonide 9mg by mouth in three daily divided doses, FK with an initial target trough level of no greater than 5-6ng/mL, and MMF (I-ISP); or (2) S-ISP including prednisone, calcineurin antagonist, and MMF. After randomization, subjects will be followed for a total of 52 weeks and assessed for adequacy of graft function, and complications of therapy, particularly ACR

ELIGIBILITY:
Inclusion Criteria: Adult patients age 18 years or older who undergo initial single-organ living- or deceased-donor liver-transplant surgery. Research participants are required to have satisfactory post-operative recovery of graft function and no post-operative renal-replacement therapy prior to starting medication according to protocol. They must also be able to take oral medications.

-

Exclusion Criteria: Patients will be excluded from the study if they are: (1) undergoing retransplantation; (2) have fulminant hepatic failure as an indication for liver transplantation; (3) have surgical complication(s) potentially affecting post-operative graft function (i.e., hepatic artery thrombosis); or have delayed initial recovery of graft function (primary non-function) requiring non-standard induction therapy. Furthermore, patients with a contraindication to budesonide (i.e., hypersensitivity) will not be included in the study

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Acute cellular rejection (ACR) | 12 months
  Incidence of ACR in budesonide treatment arm as compared to standard treatment arm

SECONDARY OUTCOMES:
Tacrolimus trough levels | 12 months
  Cumulative average trough level of tacrolimus in budesonide and standard treatment arms
Diabetes | 12 months
  Incidence of diabetes in in budesonide and standard treatment arms
Worsening kidney function | 12 months
  Incidence of worsening kidney function in budesonide and standard treatment arms
Hyptertension | 12 months
  Incidence of hypertension in in budesonide and standard treatment arms
Graft survival | 12 months
  Graft survival in budesonide and standard treatment arms
Patient survival | 12 months
  Patient survival in budesonide and standard treatment arms
Infection | 12 months
  Incidence of infection in budesonide and standard treatment arms

IPD SHARING:
Plan to Share IPD: Undecided
Annonymous IPD will be shared in the event that the study protocol is approved at other transplanting institutions who then collaborate in this study. IPD will include standard clinical and laboratory data monitored after liver transplantation

REFERENCES:
- [Background] Jonsson G, Astrom A, Andersson P. Budesonide is metabolized by cytochrome P450 3A (CYP3A) enzymes in human liver. Drug Metab Dispos. 1995 Jan;23(1):137-42. PMID 7720517
- [Background] Weber T, Kalbhenn T, Herrmann G, Hanisch E. Local immunosuppression with budesonide after liver transplantation in the rat: a preliminary histomorphological analysis. Transplantation. 1997 Sep 15;64(5):705-8. doi: 10.1097/00007890-199709150-00007. PMID 9311706
- [Background] Ozcay N, Fryer J, Grant D, Freeman D, Garcia B, Zhong R. Budesonide, a locally acting steroid, prevents graft rejection in a rat model of intestinal transplantation. Transplantation. 1997 May 15;63(9):1220-5. doi: 10.1097/00007890-199705150-00006. PMID 9158013
- [Background] Bhat M, Ghali P, Wong P, Marcus V, Michel R, Cantarovich M, Metrakos P, Deschenes M. Immunosuppression with budesonide for liver transplant recipients with severe infections. Liver Transpl. 2012 Feb;18(2):262-3. doi: 10.1002/lt.22453. No abstract available. PMID 22006869
- [Background] Lichtenstein GR, Travis S, Danese S, D'Haens G, Moro L, Jones R, Huang M, Ballard ED, Bagin R, Hardiman Y, Collazo R, Sandborn WJ. Budesonide MMX for the Induction of Remission of Mild to Moderate Ulcerative Colitis: A Pooled Safety Analysis. J Crohns Colitis. 2015 Sep;9(9):738-46. doi: 10.1093/ecco-jcc/jjv101. Epub 2015 Jun 20. PMID 26094251
- [Result] Manns MP, Woynarowski M, Kreisel W, Lurie Y, Rust C, Zuckerman E, Bahr MJ, Gunther R, Hultcrantz RW, Spengler U, Lohse AW, Szalay F, Farkkila M, Prols M, Strassburg CP; European AIH-BUC-Study Group. Budesonide induces remission more effectively than prednisone in a controlled trial of patients with autoimmune hepatitis. Gastroenterology. 2010 Oct;139(4):1198-206. doi: 10.1053/j.gastro.2010.06.046. Epub 2010 Jun 22. PMID 20600032